CLINICAL TRIAL: NCT02145988
Title: Improvement of Ankle-Brachial Index by DLBS1033 Treatment in Diabetic Patients With Peripheral Arterial Disease
Brief Title: DLBS1033 Treatment in Diabetic With Peripheral Arterial Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruitment rate is unexpectedly too low (insufficient number of eligible patients).
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS1033-0312
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Diabetes; Peripheral Arterial Disease
Keywords: DLBS1033; Peripheral arterial disease; Ankle-brachial index
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Arterial Disease | interventions — DLBS 1033

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DLBS1033 (Experimental): DLBS1033 tablet is administered at the dose of 490 mg, one tablet three times daily, every day for twelve weeks of study period
  Interventions: Drug: DLBS1033
- Placebo (Placebo Comparator): Placebo tablet is administered one tablet three times daily, every day for twelve weeks of study period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DLBS1033 — Investigational drug or placebo will be given in addition to the standard therapy: aspirin at the dose of 80 mg, once daily, every day for twelve weeks of study period
  Other Names: Disolf
  Arms: DLBS1033
Drug: Placebo — Investigational drug or placebo will be given in addition to the standard therapy: aspirin at the dose of 80 mg, once daily, every day for twelve weeks of study period
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind, double-dummy, and controlled study of DLBS1033 for the improvement of ankle-brachial index in diabetic patients with peripheral arterial disease (PAD). It is hypothesized that the addition of DLBS1033 on top of aspirin treatment will augment significantly the resting ABI in diabetes patient with PAD in comparison with that of aspirin alone.

DETAILED DESCRIPTION:
Subjects in this study will be screened consecutively and eligible subjects will be randomized to receive aspirin tablet 80 mg once daily and either the investigational drug (DLBS1033 tablet 490 mg three times daily) or its placebo, for 12 weeks.

Diabetic subjects who have been being under therapy with aspirin can directly start with study treatment. For those who are currently not under therapy with aspirin, there will be a run-in period during which they will receive (or be switched to) aspirin treatment, for two weeks. After then, they will receive study medication.

Clinical and laboratory examinations to evaluate the investigational drug's efficacy and safety will be performed at baseline and at the interval of six weeks over the twelve week-course of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any trial related activities.
* Male or female subjects of 40 - 65 years of age.
* Diagnosis of diabetes mellitus defined as HbA1c level of ≥ 6.5% (for newly diagnosed diabetes) or based on medical history.
* Presence of peripheral arterial disease with resting ankle-brachial index (ABI) of 0.41-0.90 inclusive

Exclusion Criteria:

* Females of childbearing potential: pregnancy, breast-feeding, and the intention of becoming pregnant.
* Recent stroke attack, myocardial infarction/unstable angina/acute coronary syndrome, coronary artery bypass surgery (CABG) or percutaneous transluminal coronary angioplasty (PTCA)/stent within 3 (three) months prior to screening.
* Impaired liver function: serum ALT > 2.5 times upper limit of normal.
* Impaired renal function: serum creatinine ≥ 1.5 times upper limit of normal.
* Concomitant use of other antithrombosis drugs or any antiplatelets other than the study medication.
* Subjects with concurrent herbal (alternative) medicines or food supplements
* Subjects with any other disease state, including chronic or acute systemic infections, uncontrolled illnesses or other chronic diseases, which judged by the investigator, could interfere with trial participation or trial evaluation.
* Subjects with high risk of bleeding:
* Subjects with prior experience with DLBS1033 or other oral lumbrokinase products.
* Subjects with known or suspected allergy to any of study medications used in the study, including other lumbrokinase products.
* Subjects with known or suspected allergy or resistant to aspirin.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Resting ankle-brachial index (ABI) | Week 0 and 12
  The change of resting ABI

SECONDARY OUTCOMES:
Resting ABI | Week 0 and 6
  The change of resting ABI
hs-CRP | Week 0, 6, and 12
  The change of hs-CRP
Thromboxane B2 | Week 0, 6, and 12
  The change of thromboxane B2
Fibrinogen | Week 0, 6, and 12
  The change of fibrinogen
d-dimer | Week 0, 6, and 12
  The change of d-dimer
Routine hematology | Week 0, 6, and 12
  Routine hematology measured includes: hemoglobin, hematocrit, RBC, WBC, differentiation of WBC, and platelet count
Liver function | Week 0 and 12
  Liver function measured includes: serum ALT, AST, and alkaline phosphatase
Renal function | Week 0 and 12
  Renal function measured includes: serum creatinine and blood urea nitrogen (BUN)
Haemostasis parameters | Week 0, 6, and 12
  Haemostasis parameters measured includes: prothrombin time (PT) and activated partial thromboplastin time (aPTT)
Adverse events | Week 0 - 12
  Adverse events, including bleeding events, will be observed and carefully evaluated along the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ketut Suastika, Prof, SpPD, MD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, University of Udayana/Sanglah Hospital
Locations (2):
- Indonesia (2):
  - Department of Internal Medicine, Faculty of Medicine, University of Udayana/Sanglah Hospital, Denpasar, Bali
  - Department of Internal Medicine, RSUD Wangaya, Denpasar, Bali